CLINICAL TRIAL: NCT03281928
Title: Effect of Dietary Sodium and Potassium Citrate on Renal Mineral Handling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to IRB expiration. A new protocol (IRB22-1817) was submitted to continue the research.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB17-0992
Record Dates: First submitted 2017-09-08; First posted 2017-09-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Sodium; Potassium Citrate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Sodium plus Potassium Citrate (Experimental)
  Interventions: Dietary Supplement: Sodium and Potassium Citrate
- Low Sodium plus placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- High Sodium plus Potassium Citrate (Experimental)
  Interventions: Dietary Supplement: Sodium and Potassium Citrate
- High Sodium plus placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium and Potassium Citrate — Sodium and potassium citrate levels will be altered in diet and renal mineral handling will be measured as compared to placebo.
  Arms: High Sodium plus Potassium Citrate; Low Sodium plus Potassium Citrate
Dietary Supplement: Placebo — Sodium without Potassium Citrate
  Arms: High Sodium plus placebo; Low Sodium plus placebo

SUMMARY:
This study intends to characterize the affect of sodium and potassium citrate in the diet on renal function.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 70, approximately equal numbers of men and women
* studied by endoscopy with complete papillary mapping and grading
* stone formers

Exclusion Criteria:

* Patients with primary renal diseases or renal impairment (eGFR < 90), or medical conditions such as diabetes, or systemic diseases or medications that alter calcium metabolism
* Patients with known bladder voiding problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Urine Calcium levels | 10 days
  Amount of calcium in the urine will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States